CLINICAL TRIAL: NCT04648982
Title: Psychiatric Inpatient Discharge Data - Rwanda
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: University of Rwanda (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AUUR2020DKRW_2
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-11

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Admission to inpatient psychiatric unit — All persons in the study are hospitalized at the only inpatient mental health hospital in Rwanda - Ndera. Data will be collected when the person is being discharged.

SUMMARY:
The aim is to provide a comprehensive assessment regarding the service provision and the accessibility to intensive mental health care in Rwanda

DETAILED DESCRIPTION:
For a one-year period, descriptive data on all inpatients with age > 18 years, discharged from Ndera Hospital the only inpatient psychiatric hospital in Rwanda, will be collected from files. The descriptive data includes diagnosis, duration of hospitalization, medication, addiction, insurance, Somatic- and psychiatric comorbidity, referral pathways, employment status, number of previous hospitalizations. To the investigators' knowledge, there is no descriptive data on psychiatric inpatients in the country of Rwanda. Therefore, this. Information will be crucial for understanding the service provision at the referral hospitals and the accessibility to intensive mental health care in Rwanda. The data will be anonymized and recorded - this ensures the data cannot be linked to anyone subject which supplied it.

ELIGIBILITY:
Inclusion Criteria:

* All patients discharged from the inpatient psychiatric unit at Ndera Hospital, Rwanda

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons that are hospitalized due to mental health concerns in Rwanda.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis | 1 year
  Data will be collected from files
Psychiatric comorbidity | 1 year
  Data will be collected from files
Somatic comorbidity | 1 year
  Data will be collected from files
Alcohol or drug addiction | 1 year
  Data will be collected from files
Medical drug provided during this hospitalisation | 1 year
  Data will be collected from files
Who made the referral | 1 year
  Data will be collected from files
Number of previous hospitalisations | 1 year
  Data will be collected from files
Insurance | 1 year
  Data will be collected from files

CONTACTS AND LOCATIONS:
Overall Officials: Per Kallestrup, Prof., Study Chair — University of Aarhus
Locations (2):
- Rwanda (2):
  - Ndera Hospital, Huye
  - Ndera Hospital, Kigali

IPD SHARING:
Plan to Share IPD: No